CLINICAL TRIAL: NCT07166744
Title: Contribution of Pathological Alpha-Synuclein as a Diagnostic Biomarker for Dementia With Lewy Bodies
Acronym: QuIC-Lewy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9047
Record Dates: First submitted 2025-08-01; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Dementia With Lewy Bodies (DLB); Alzheimer's Disease (AD)
MeSH Terms: conditions — Lewy Body Disease; Alzheimer Disease | interventions — Functional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Disease/dementia with lewy Bodies (DLB) (Experimental): Disease/Dementia with lewy bodies(DLB) according to the criteria of McKeith et al. 2017 and 2020, + positive DAT-scan at inclusion applying, if necessary, usual biomarkers such as polysomnography and MIBG scintigraphy. Patients with non-significant (0 or 1 out of 3) Alzheimer's disease LCS biomarkers (P-Tau, Tau, and Abeta42/40) will be considered as true MCL following lumbar puncture as part of the protocol.
  * Biological : blood sampling, nasopharyngeal swab
  * Procedure : Lumbar puncture
  * Behavioral : clinical, functional, cognitive and psychiatric evaluations
  * Other : MRI
  Interventions: Other: Biological : blood sampling; Other: nasopharyngeal swab; Other: Procedure : Lumbar puncture; Other: Behavioral : clinical, functional, cognitive and psychiatric evaluations; Other: MRI
- Alzheimer's disease arm (Active Comparator): Alzheimer's disease (AD) according to the criteria of Dubois et al., 2014.
  * Biological : blood sampling, nasopharyngeal swab
  * Procedure : Lumbar puncture
  * Behavioral : clinical, functional, cognitive and psychiatric evaluations Other : MRI
  Interventions: Other: Biological : blood sampling; Other: nasopharyngeal swab; Other: Procedure : Lumbar puncture; Other: Behavioral : clinical, functional, cognitive and psychiatric evaluations; Other: MRI
- Fronto-temporal diseases arm (Active Comparator): Fronto-temporal disease (FTD) in the broad sense: taupathy or tardopathy: fronto-temporal lobar dementia (FTLD) according to the criteria of Rascovsky et al., 2011, or cortico-basal degeneration (CBD) according to the criteria of Amstrong et al., 2013, or supranuclear palsy according to the criteria of Höglinger et al., 2017, or Limbic-predominant age-related TDP-43 encephalopathy (LATE).
  * Biological : blood sampling, nasopharyngeal swab
  * Procedure : Lumbar puncture
  * Behavioral : clinical, functional, cognitive and psychiatric evaluations Other : MRI
  Interventions: Other: Biological : blood sampling; Other: nasopharyngeal swab; Other: Procedure : Lumbar puncture; Other: Behavioral : clinical, functional, cognitive and psychiatric evaluations; Other: MRI
- Psychiatric disorders arm (Active Comparator): Psychiatric disorders such as depression, bipolarity or schizophrenia, etc according to DSM 5 criteria.
  * Biological : blood sampling, nasopharyngeal swab
  * Procedure : Lumbar puncture
  * Behavioral : clinical, functional, cognitive and psychiatric evaluations Other : MRI
  Interventions: Other: Biological : blood sampling; Other: nasopharyngeal swab; Other: Procedure : Lumbar puncture; Other: Behavioral : clinical, functional, cognitive and psychiatric evaluations; Other: MRI

INTERVENTIONS:
Other: Biological : blood sampling — will be collected from the patient
Other: nasopharyngeal swab — will be collected from the patient
Other: Procedure : Lumbar puncture — will be collected from the patient
Other: Behavioral : clinical, functional, cognitive and psychiatric evaluations — will be collected from the patient
Other: MRI — will be done on the patient

SUMMARY:
Alzheimer's disease and dementia with Lewy bodies (DLB) are the two main age-related neurodegenerative cognitive disorders. Differential diagnosis between these conditions is challenging, both at the prodromal and dementia stages. The lack of a precise diagnosis can be particularly harmful for patients with DLB, as up to 80% of them show severe adverse reactions to antipsychotic medications, including falls, confusion, and even death. The diagnosis of Alzheimer's disease has improved with cerebrospinal fluid (CSF) biomarkers such as Tau, phosphorylated Tau (P-Tau), and the Aβ42/Aβ40 ratio (Lehmann et al., 2018). However, differentiating Alzheimer's disease from DLB remains difficult: 1 to 3 Alzheimer's biomarkers are frequently positive in the CSF of patients with DLB: in 49% of cases at the prodromal stage and up to 72% at the dementia stage. Moreover, total α-synuclein measurement in CSF has not proven to be diagnostically reliable. The DAT-scan, sometimes used as a supportive tool, is an expensive technique and lacks sensitivity, with detection rates of only 78% in dementia-stage DLB and 54% in prodromal DLB.

Given these limitations, identifying specific biomarkers for DLB, particularly pathological α-synuclein, is a critical objective. α-synuclein is the main protein component of Lewy bodies, whose abnormal β-sheet conformation promotes aggregation and prion-like propagation. Conventional measurements of total α-synuclein in CSF have failed to achieve sufficient diagnostic specificity. In contrast, detecting aggregated or pathological forms of α-synuclein in CSF appears to be a promising approach for improving the diagnosis of synucleinopathies. New techniques based on α-synuclein aggregation amplification have shown encouraging results in retrospective studies including neuropathologically confirmed cases (Bargar et al., 2021; Rossi et al., 2020). However, prospective evaluation of these methods in real-world clinical settings is still lacking. We hypothesize that a specific assay targeting pathological α-synuclein in CSF could reliably distinguish patients with DLB from those with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* - Patient, male or female, age equal or over 50 with signs suggestive of one of the following conditions: Lewy body disease (LBD) according to the criteria of McKeith et al. 2017 and 2020, + positive DAT-scan at inclusion applying, if necessary, usual biomarkers such as polysomnography and MIBG scintigraphy. Patients with non-significant (0 or 1 out of 3) Alzheimer's disease LCS biomarkers (P-Tau, Tau, and Abeta42/40) or Alzheimer's disease (AD) biomarkers (0 or 1 out of 3) will be considered as true MCL following lumbar puncture as part of the protocol.
* Alzheimer's disease (AD) according to the criteria of Dubois et al. 2014, or
* MCL + AD disease according to the criteria of McKeith et al. 2017 and 2020 + a positive DAT-scan at inclusion and Dubois et al. 2014, or
* Fronto-temporal diseases (FTD) in the broad sense: taupathy or tardopathy: fronto-temporal lobar dementia (FTLD) according to the criteria of Rascovsky et al., 2011, or cortico-basal degeneration (CBD) according to the criteria of Amstrong et al., 2013, or supranuclear palsy according to the criteria of Höglinger et al., 2017, or age-related predominantly limbic TDP-43 encephalopathy (LATE).
* Psychiatric disorders such as depression, bipolarity, schizophrenia according to DSM 5 criteria.
* Patient accompanied by a caregiver or a person likely to provide information about him/her (interview, telephone contact) in case the investigator deems the patient unable to provide this information alone.
* Patient able to understand the aims and risks of the research and to give dated, signed informed consent (or consent given by the trusted support person/guardian, or in the presence of the curator if the patient is under guardianship or curatorship).
* Patient affiliated to a social health insurance protection.
* Patient presenting at syndromic level :

either mild cognitive impairment (according to Petersen criteria) or mild, moderate or severe dementia (MMSE 30 to 5 included)

Exclusion Criteria:

* Patient with other neurological disease including, but not limited to, the following conditions: cerebral tumor, cerebrovascular accident with cognitive impairment, multisystem atrophy, etc, as judged by the investigator.
* Patient with a contraindication to lumbar puncture.
* Patient with a contraindication to cerebral MRI (patients included in Strasbourg only).
* Any reason making it impossible to follow up the patient during the study period (planned move, etc.).
* Patient under Legal safeguard ("sauvegarde de justice")- Impossibility of giving the patient informed information (patient in emergency or life-threatening situation).

Patients under guardianship or curatorship may be included in the study; in fact, in severe to moderately severe patients (MMS<15), such a measure is often in place.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic value of pathological α-synuclein in cerebrospinal fluid (CSF) using lumbar puncture. | Day 0
  Pathological alpha-synuclein aggregation and amplification will be measured through its binding with fluorescent Thioflavin T. Fluorescence will be measured as a percentage using a spectrophotometer.

IPD SHARING:
Plan to Share IPD: No